CLINICAL TRIAL: NCT06745375
Title: Evaluation of the Vision and Fit of Commercially Available Correct Powered (Prescription) Contact Lenses Compared to Lenses Within a Range of ± 2.00 Dioptres (Strength/Power of Lens) From the Prescription
Brief Title: Assessment of the Relationship of Soft Contact Lens Fit and Power (Fit & Lens pOwer Soft lenSes)
Acronym: FLOSS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Aston University (Other)
Collaborators: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HLS21201
Record Dates: First submitted 2024-12-09; First posted 2024-12-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants Study; Contact Lens Wear; Contact Lens Fit
Keywords: contact lens; contact lens wear; contact lens fit
MeSH Terms: interventions — Contact Lenses, Extended-Wear

STUDY DESIGN:
Intervention Model Description: This crossover study compares patients' actual prescription contact lenses with lenses ±2.00 dioptres to assess differences in fit. Key fitting metrics include lens movement (<1.00 mm), coverage, and push-up tests. Using G*Power (v3.1.9.4), a sample size of 38 was calculated. The study uses paired assessments (same participant wears both lenses) to evaluate lens movement in mm. Literature reports mean ± SD of 0.352 ± 0.355 mm and 0.269 ± 0.179 mm, with high correlation (r = 0.95) (Belda-Salmerón et al.). A clinically significant difference is set at 0.25 mm. To achieve 80% power with a 5% Type I error and accounting for a 10% dropout rate, 38 participants are required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy participants (Experimental): All healthy participants wear two different contact lenses, one with the correct power and one with +/- 2.00 Ds to actual refraction. All lenses are commercially available. No 2nd arm.
  Interventions: Device: contact lens wear

INTERVENTIONS:
Device: contact lens wear — participants wear two different powered contact lenses (one with actual power, and one +/- 2.00Ds) contact lenses. No 2nd arm

SUMMARY:
The purpose of this study is to evaluate whether altering the optical power (in dioptres) of a contact lens affects both vision and lens fit. As the majority of modern contact lens wearers prefer daily disposable soft lenses, the trial lenses used in this study-provided by CooperVision-reflect this trend, representing nearly 80% of the current UK market.

This study aims to generate data supporting the use of contact lenses with powers that do not precisely match a participant's visual prescription (within ±2.00 dioptres) as a viable temporary alternative when the exact required power is unavailable.

At present, there is no published literature in the context of modern contact lens design that compares the fitting characteristics of 'fit-for-purpose' lenses with those of lenses from the same design family that would not typically be selected due to power mismatch.

DETAILED DESCRIPTION:
This study aims to evaluate the vision and fit of commercially available prescription contact lenses of different strengths to determine whether this affects the final lens selection and, if so, how. In addition, the study will compare subjective comfort and key fitting criteria such as centration, movement, tightness, coverage, and overall impression.

These data could help eye care practitioners use lenses they already have in stock instead of ordering new ones and requiring patients to return. Understanding whether these lenses fit similarly could make the process more convenient for both patients and practitioners. Patients would receive their lenses more quickly, and eye care providers could manage their existing stock more effectively.

The two visits will take place at the Aston University Eye Clinic. Data collection and assessments will include:

Participant's age, ethnicity, sex, and ocular history to determine eligibility [recorded electronically on a secure computer].

A standardised OSDI questionnaire (paper copy only), which quantifies dry eye symptoms, severity, and frequency (e.g. in the past week, how often participants' eyes felt gritty, watery, itchy, or burning, and how many times they experienced these symptoms), will be administered at the first visit after written consent. The completed questionnaire will be scanned and uploaded to BOX.

Both Visit One and Visit Two will include:

Application of contact lenses to the participant's eyes. Lens powers will be randomised between visits for each participant.

Comfort assessment using:

A visual analogue scale (paper-based) from "most comfortable" to "least comfortable," where participants mark their comfort level.

A numerical rating (1-10) of comfort, recorded electronically. Vision assessment after lens application, both objectively (autorefractor) and subjectively, as in routine clinical practice.

A video-recorded ocular assessment of the contact lens fit, including horizontal lens movement, blink-induced movement, and lens centration.

After data collection is complete and the lenses are removed at Visit Two, participants will be asked which lenses they preferred [recorded electronically].

The data collection follows standardised contact lens assessment protocols used in both primary and secondary care optometry.

A participant's current eye care practitioner will not be informed of their participation or the corresponding assessments/data unless clinically significant findings are discovered and the participant consents to sharing this information. Participants will be informed of the lens brand and manufacturer used in the study so that, if they find the lenses more comfortable than their current ones (if applicable) or are considering contact lenses, they may discuss this with their eye care practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-60 years of age
* Vision correctable to at least 6/12 (20/40) or better in each eye
* with mental capacity to provide written consent in English (as per the Mental Capacity Act, 2005).
* happy to wear investigational contact lenses

Exclusion Criteria:

* Any active infection or inflammation, history of major systemic or ophthalmic conditions
* use of systemic or topical medications known to affect the eye in the previous 3 months
* history of ocular surgery, currently enrolled on another study/clinical trial that may impact outcome
* any other contraindications for typical contact lens wear
* As per the Mental Capacity Act, 2005, participants will be automatically excluded if not deemed to have Capacity for consent or under the age of 18.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Soft contact lens movement: Subjective and objective assessment of soft contact lens movement. | within 30 mins of lens wear
  Lens movements will be graded between 0.25 - 0.50 mm = Optimum, <0.25 = Less movement; >0.50mm is more movement.
Soft contact lens horizontal lag:Subjective and objective assessment of soft contact lens lag. | within 30 mins of lens wear
  Lens lag will be graded as: <50% lag = less leg, 50% to 100% is optimum lag, >100% = high lag.
Soft contact lens tightness: graded subjectively as optimum, loose and tight | within 30 mins of lens wear
  Soft contac tlens tightness

SECONDARY OUTCOMES:
Assessment of ocular comfort with soft contact lenses | within 30 mins of lens wear
  Ocular comfort is graded by particpants 1-10 (1 being very uncomfortable and 10 being highly comfortable)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Optometry, Aston Eye Clinic, Birmingham, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This has not been planned, yet but there is no reason cant be done by the end of study.